CLINICAL TRIAL: NCT06791681
Title: Clinical Study for Evaluating ESO-T01 Injection's Safety and Efficacy in Treating Relapsed/refractory Multiple Myeloma
Brief Title: A Study of ESO-T01 in Treating Relapsed/ Refractory Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chunrui Li (Other)
Collaborators: Shenzhen Pregene Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chunrui Li, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG2402E
Record Dates: First submitted 2025-01-09; First posted 2025-01-24 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-11

CONDITIONS: Relapsed/ Refractory Multiple Myeloma
Keywords: ESO-T01; Multiple Myeloma; in vivo
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ESO-T01 treatment group (Experimental): the third-generation self-inactivating lentiviral vector
  Interventions: Drug: ESO-T01

INTERVENTIONS:
Drug: ESO-T01 — ESO-T01 injection is the third-generation self-inactivating lentiviral vector targeting T cells in vivo, which carries a single VHH-directed BCMA-targeted CAR.
  Other Names: BCMA CAR-T

SUMMARY:
This is a single center, single arm, open-label, dose-escalation clinical study to observe the safety, tolerability, preliminary efficacy, pharmacokinetics, pharmacodynamics of ESO-T01 injection for treating patients with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
ESO-T01 injection is the third-generation self-inactivating lentiviral vector targeting T cells in vivo, which carries a single VHH-directed BCMA-targeted CAR. Before infusion, the patients will be given the prophylaxis of acetaminophen and diphenhydramine. The designed dose-escalation includes four dose groups of dose A, B, C, and D. After infusion, patients will be followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years；
2. Diagnosis of multiple myeloma (MM) confirmed according to the IMWG diagnostic criteria, with BCMA expression on MM cells determined by flow cytometry or immunohistochemistry;
3. Previously treated with at least 2 lines of anti-MM therapy, with at least 1 complete treatment cycle for each line, and disease progression within 12 months after the most recent anti-myeloma treatment, or being refractory to both immunomodulatory drugs and proteasome inhibitors, along with disease progression within 2 months after the most recent anti-myeloma treatment (according to the IMWG diagnostic criteria);
4. Disease must be measurable at screening, meeting at least one of the following criteria:Serum M-protein level ≥ 0.5 g/dL; Urinary M-protein level ≥ 200 mg/24h; Serum involved free light chain ≥ 10 mg/dL and an abnormal serum free light chain κ/λ ratio;
5. ECOG score 0-2, with an expected survival time ≥ 3 months;
6. Bone marrow function at screening (or within 2 months prior to screening) meets the following criteria: a.Hemoglobin ≥ 6 g/dL (no red blood cell transfusion within 1 week before screening), recombinant human erythropoietin is allowed; for patients who meet the ≥6 g/dL criterion at screening, red blood cell transfusion is allowed to maintain hemoglobin ≥ 6 g/dL; b.Absolute neutrophil count (ANC) ≥ 600/μL (no use of granulocyte colony-stimulating factor (G-CSF) within 1 week or pegylated G-CSF within 2 weeks prior to screening); c. Platelet count ≥ 50,000/μL; d. Lymphocyte count ≥ 500/μL; e. Absolute CD3-positive T cell count ≥ 150/μL;
7. Renal function at screening (or within 2 months prior to screening) should be normal, with a creatinine clearance ≥ 45 mL/min;
8. Liver function at screening (or within 2 months prior to screening) must meet the following criteria: a. Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 3.0 × the upper limit of normal (ULN); b. Total bilirubin (TBIL) and alkaline phosphatase (AKP or ALP) ≤ 2.0 × ULN (except for congenital hyperbilirubinemia, such as Gilbert's syndrome, where direct bilirubin can be ≤ 1.5 × ULN); c. Albumin ≥ 3 g/dL;
9. Cardiac function at screening (or within 2 months prior to screening) must meet the following criteria: a. Left ventricular ejection fraction ≥ 40% (measured by echocardiogram or MUGA scan); b. No clinically significant pericardial effusion detected; c. No clinically significant ECG abnormalities detected;
10. Pulmonary function at screening (or within 2 months prior to screening) must meet the following criteria: Oxygen saturation ≥ 90%;No clinically significant pleural effusion detected;
11. For women of childbearing potential, a negative pregnancy test must be obtained at screening and prior to drug infusion, and they must not be breastfeeding;
12. Male and female subjects of childbearing potential must agree to use effective contraception from the time of informed consent until 1 year after the study drug administration;
13. Male and female subjects of childbearing potential must agree not to donate sperm or eggs (oocytes) or other reproductive cells from the time of informed consent until 1 year after the study drug administration;
14. The participant or their legally authorized representative must provide written informed consent (ICF), indicating their understanding of the purpose and procedures of the study and their willingness to participate.

Exclusion Criteria:

1. Previous anticancer treatment (as determined by the investigator): a. Received targeted therapy, epigenetic therapy, other investigational drugs, or treatment using invasive investigational medical devices within 5 half-lives; b. Received immune/non-immune-directed systemic therapy within 1 week; Received cytotoxic therapy within 1 week; c. Received proteasome inhibitors or immunomodulatory agent therapy within 2 weeks; d. Received radiotherapy within 4 weeks (if the radiation field covered ≤5% of bone marrow reserve, the subject is eligible regardless of the date of radiotherapy completion);
2. Received allogeneic HSCT within 6 months prior to infusion, or autologous HSCT within 3 months prior to infusion;
3. Other malignancies prior to screening (except the following): Malignancies treated with curative intent and no evidence of active disease ≥2 years before enrollment; Adequately treated non-melanoma skin cancer with no evidence of disease;
4. Previously treated with any viral therapy using VSVG pseudotype virus;
5. Serious uncontrolled infections during screening: Bacterial, viral, fungal, etc. infections;
6. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with elevated peripheral blood HBV DNA levels within 6 months prior to infusion; Positive for hepatitis C antibody (HCV Ab) with elevated peripheral blood HCV RNA levels; Positive for HIV antibody; Positive for syphilis;
7. Symptomatic heart failure or significant arrhythmias: NYHA Class III or IV congestive heart failure; Myocardial infarction or coronary artery bypass grafting (CABG) or coronary stent implantation within ≤6 months prior to signing ICF; Clinically significant ventricular arrhythmias or unexplained syncope (except when caused by vasovagal or dehydration); Significant non-ischemic cardiomyopathy history;
8. Other significant diseases: Primary immunodeficiency; Stroke or seizure within 6 months prior to screening; Obvious clinical evidence of dementia or altered mental status; History of Parkinson's disease or Parkinsonism;
9. Surgery within 2 weeks prior to treatment or planned surgery within 2 weeks post-treatment, except for local anesthesia procedures;
10. Use of live-attenuated vaccines within 1 month before treatment;
11. Known severe allergic reaction to ESO-T01 or its formulation components;
12. Known severe allergic reaction to Tocilizumab;
13. Inability to establish venous access;
14. Any other condition deemed by the investigator as unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Dose-limiting toxicities (DLTs) are evaluated between the infusion and 28 days post-infusion.
  Dose limiting toxicity will be assessed after injection
Cytokine release syndrome (CRS) | up to Day 28 post-infusion
  Cytokine release syndrome (CRS) would be graded according to the ASTCT consensus.
immune cell-associated immune effector cell-associated neurotoxicity syndrome (ICANS) | up to Day 28 post-infusion
  ICANS would be scored according to Immune Effector Cell-Associated Encephalopathy (ICE), and then graded by the ASTCT consensus.
Treatment-associated adverse effects (AEs) | up to 2 years after treatment of ESO-T01
  All other AEs would be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
Overall response rate (ORR) | Day 14, Day 28, Month 2 , Month 3, Month 6, Month 9, Month 12, Month 18, Month24 after the treatment of ESO-T01.
  Clinical efficacy can be evaluated according to the 2016 International Myeloma Working Group consensus criteria.
Complete response (CR) rate | Day 14, Day 28, Month 2 , Month 3, Month 6, Month 9, Month 12, Month 18, Month24 after the treatment of ESO-T01.
  sCR/CR can be evaluated according to the 2016 International Myeloma Working Group consensus criteria.
Duration of response (DOR) | Through study completion, an average of 2 year
  DOR is defined as the interval between the first sCR, CR, VGPR, or PR after infusion and the disease progression or death.
Progression-free survival (PFS) | up to 2 years after treatment of ESO-T01.
  PFS is defined as the interval between a subject's receipt of ESO-T01 infusion and the first assessment of disease progression or death.
Overall survival (OS) | up to 2 years after treatment of ESO-T01
  OS is defined as the interval between a subject's receipt of ESO-T01 infusion and death from any cause.
Cmax | Baseline, Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 14, Day 17, Day 21, Day 24, Day 28, Month 2 , Month 3, Month 6, Month 9, Month 12, Month 18, Month24 after the treatment of ESO-T01
  CAR-T kinetics would be detected by flow cytometry and droplet digital PCR in peripheral blood and bone marrow at each important time points. Cmax is the peak expansion value of CAR-T cells.
Tmax | Baseline, Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 14, Day 17, Day 21, Day 24, Day 28, Month 2 , Month 3, Month 6, Month 9, Month 12, Month 18, Month24 after the treatment of ESO-T01
  CAR-T kinetics would be detected by flow cytometry and droplet digital PCR in peripheral blood and bone marrow at each important time points. Tmax is the time of the occurrence of expansion peak.
AUC(0-day 28) | Baseline, Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 14, Day 17, Day 21, Day 24, Day 28 after the treatment of ESO-T01
  CAR-T kinetics would be detected by flow cytometry and droplet digital PCR in peripheral blood and bone marrow at each important time points. Cmax is the peak expansion value of CAR-T cells. AUC(0- day28) refers to the area under curve of CAR-T cell expansion between infusion and day 28 post infusion. They all reflect the pharmacokinetics.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: January 2026-unending